CLINICAL TRIAL: NCT00737607
Title: Clinical Study of Microendoscopic Decompressive Laminotomy for Treatment of Lumbar Spinal Stenosis
Brief Title: Clinical Outcome Study of Minimally Invasive Decompression for Lumbar Spinal Stenosis
Acronym: MEDLLSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Jwo-Luen Pao, Far-Eastern Memorial Hospital
Other Study IDs: 97034; FEMH-96-C-039
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Lumbar Spinal Stenosis
Keywords: outcome; surgery; lumbar spinal stenosis; minimally invasive
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a prospective outcome study to evaluate the effectiveness and treatment outcomes of microendoscopic decompressive laminotomy (MEDL) with objective evaluation tools. The patients who fulfill the selection criteria will be enrolled to collect the pre-operative clinical data including demographic data, image studies, and functional evaluation for neurological symptoms and disability.

The patient will receive MEDL and post-operative follow-up will be arranged at 1 week, 1 month, 6 months, and 12 months after the operation. All the collected data will be analyzed to evaluate the efficacy and treatment results of MEDL.

DETAILED DESCRIPTION:
The patients undergoing microendoscopic decompressive laminotomy (MEDL) for lumbar spinal stenosis (LSS) between will be enrolled in this prospective study. The patients included must fulfill the following selection criteria:

* neurogenic claudication or radicular leg pain with associated neurologic signs referring to the LSS syndrome;
* moderate to severe spinal canal stenosis shown on cross-sectional imaging such as MRI or CT scan;
* failure of conservative treatment for at least three months.

The patients who presents with either mechanical low back pain or segmental instability. Mechanical lower back pain is defined as pain that was induced by posture change, or that prevents the patient from sitting or standing for more than 30 minutes. Patients are considered to have segmental instability if they had isthmic spondylolisthesis, degenerative spondylolisthesis with more than 4 mm of translation or intervertebral angle reversal on dynamic radiographs.18 Surgical techniques

All the surgical procedures will be performed by a single surgeon (J. P.). The patients is positioned prone on the Relton-Hall frame after general anesthesia. Decompression is done under the endoscope with the tubular retraction system METRx (Medtronics, Minneapolis, MN). For patients with unilateral neurological symptoms, we will perform unilateral laminotomy and foraminotomy. For patients with bilateral neurological symptoms, we will performe unilateral laminotomy for bilateral decompression (ULBD) to decompress the central canal and bilateral lateral recesses.

When performing multiple-level decompression, the skin incision will be centered at the midpoint between selected intervertebral disc levels. The incision can be mobilized one level above or below after releasing the underlying connective tissues. Then we can set up the tubular retractor system through separate muscular portals for each level. For patients with small stature, we can perform a three-level surgery through a single surgical wound, just as the same size as we perform the single-level surgery.

All the patients will have routine AP, lateral, dynamic lateral radiographs pre-operatively, six months after the surgery, and at final follow-up. Post-operative instability is defined as progression of listhesis or scoliosis on dynamic radiographs.

Every patient will MR images of the lumbar spine before the surgery. The severity of stenosis is classified according to the cross sectional area of the dura sac at the axial plane on T1-weighted MR images-severe stenosis for less than 76 mm2, moderate stenosis for between 76 and 100 mm2, and mild stenosis for more than 100 mm2. When MRI is contraindicated, CT-myelography will be used instead.

Outcomes assessment will done with Oswestry Disability Index (ODI) for the overall disability and the Japanese Orthopedic Association (JOA) score for the clinical symptoms and signs. The patients will receive evaluation before the surgery, at six months, and at the final follow-up examination. The range of ODI is 100 ~ 0 with a lower index corresponding to a better result. Significant improvement is defined as more than 15 points of improvement after the treatment. The range of JOA score is -3 ~ 29 with a higher score corresponding to a better result. The improvement rate based on JOA score is calculated as follows: (pre-operative score - post-operative score)/(29 - pre-operative score) × 100%. The clinical results are classified into four grades by the improvement rate: excellent (more than 75%), good (between 51% and 75%), fair (between 26% and 50%), and poor (less than 26%). The success of treatment is defined as more than 25% improvement rate in JOA score.20 At the final follow-up, we will inquire each patient if he or she is satisfied with the treatment results.

The data about the pre-operative comorbidities, intra-operative, peri-operative, and post-operative complications will be retrieved from medical chart review.

Distribution of gender, age, clinical characteristics (coexistence of spondylolisthesis or scoliosis, severity of stenosis, and levels of decompression), and self-assessed satisfaction by the binary outcome of treatment (success or not, based on the JOA score; significant improvement of not, base on the ODI) will be tabulated. Fisher exact test will be preformed to compare the difference between the two groups. Odds ratios will be calculated by using the univariate logistic regression. Variables with two-sided p-value less than 0.05 were considered as significant factors associated with successful treatment. All statistical analyses are performed with statistical software, SAS version 9.1 (SAS Institute Inc, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* neurogenic claudication or radicular leg pain with associated neurologic signs referring to the LSS syndrome
* moderate to severe spinal canal stenosis shown on cross-sectional imaging such as MRI or CT scan
* failure of conservative treatment for at least three months

Exclusion Criteria:

* mechanical low back pain or segmental instability

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with degenerative lumbar spinal stenosis who failed conservative treatment.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jwo-Luen Pao, MD, Principal Investigator — Far-Eastern Memorial Hospital, Taipei, Taiwan
Locations (1):
- Far-Eastern Memorial Hospital, Taipei, Taiwan